CLINICAL TRIAL: NCT05386407
Title: Telemedically Assisted Sampling of COVID-19 Patients - Is the Sampling Quality Sufficient: An Interventional Randomized Method Comparison Study
Brief Title: Telemedically Assisted Sampling of COVID-19 Patients - Is the Sampling Quality Sufficient
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Teststation Praxis Dr. med Bielecki (Other)
Responsible Party: Principal Investigator, Eisenring, Principal Investigator, Teststation Praxis Dr. med Bielecki
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2021-02508
Record Dates: First submitted 2022-05-06; First posted 2022-05-23 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Telemedicine; Pharynx; COVID-19
Keywords: Telemedicine; supervised testing; nasopharyngeal swab,; COVID-19; rapid diagnostic tests
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: interventional randomized method comparison study
Who Masked: Investigator, Outcomes Assessor
Masking Description: Our hypothesis is that, applying a strict standard operating procedure (SOP, attached), guided oropharyngeal + nasal (OP+N) self-sampling (GSS) is non-inferior to nasopharyngeal (NP) or OP+N sampling performed by health care professionals (HCP), and that guided OP+N sampling is superior to unsupervised OP+N self-sampling (USS).
  After giving informed consent by signing the consent form, patients will be randomized to either OP+N GSS - or to OP+N USS.
  After performing either procedure, they will continue to be sampled by HCP OP+N and HCP NP.
  The outcome assessors and the investigators will be blinded to the randomization to either OP+N GSS - or to OP+N US
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- telemedically assisted guided oropharyngeal + nasal (OP+N) self-sampling (GSS): OP+N GSS (Experimental): After performing the telemedically assisted OP+N GSS procedure, the patients will continue to be sampled by HCP OP+N and HCP NP.
  Interventions: Diagnostic Test: telemedically guided oropharyngeal + nasal (OP+N) self-sampling (GSS) and nasopharyngeal (NP) or OP+N sampling performed by health care professionals (HCP)
- unsupervised OP+N self-sampling (USS): OP+N USS (Experimental): Written instructions on how to perform a self-test will be provided, representing the instructions that come along with a commercially available rapid test set. An instructional online video tutorial or similar would also account as the latest state of the art.30 However, this has not yet been implemented comprehensively with all available test sets.
  After performing the OP+N USS procedure, the patients will continue to be sampled by HCP OP+N and HCP NP.
  Interventions: Diagnostic Test: telemedically guided oropharyngeal + nasal (OP+N) self-sampling (GSS) and nasopharyngeal (NP) or OP+N sampling performed by health care professionals (HCP)

INTERVENTIONS:
Diagnostic Test: telemedically guided oropharyngeal + nasal (OP+N) self-sampling (GSS) and nasopharyngeal (NP) or OP+N sampling performed by health care professionals (HCP) — After giving informed consent by signing the consent form, patients will be randomized to either OP+N GSS - or to OP+N USS.
  After performing either procedure, they will continue to be sampled by HCP OP+N and HCP NP.
  Other Names: oropharyngeal + nasal (OP+N) sampling performed by health care professionals (HCP)

SUMMARY:
The Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-COV-2) pandemic has resulted in more than 3.8 billion registered tests, 275 million positive cases, and 5 million deaths worldwide. Early and regular testing has been an important pillar of secondary prevention since the beginning.

However, this pandemic has also fostered solutions in the form of e telemedicine with enormously increased applicability.

The question of whether telemedically supervised testing with SARS-CoV-2 Rapid Antigen Tests is non-inferior to the same tests being carried out by trained personnel in test centers is still unanswered.

With this study, the investigators aim to compare and evaluate the reliability and sampling quality of telemedically guided self-performed rapid tests for professional use compared to professional sampling by healthcare personnel.

Our hypothesis is that, applying a strict standard operating procedure (SOP, attached), guided oropharyngeal + nasal (OP+N) self-sampling (GSS) is non-inferior to nasopharyngeal (NP) or OP+N sampling performed by health care professionals (HCP), and that guided OP+N sampling is superior to unsupervised OP+N self-sampling (USS).

DETAILED DESCRIPTION:
BACKGROUND AND PROJECT RATIONALE

The Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-COV-2) pandemic has resulted in more than 3.8 billion registered tests, 275 million positive cases, and 5 million deaths worldwide. Early and regular testing has been an important pillar of secondary prevention since the beginning.

However, this pandemic has also fostered solutions in the form of e telemedicine with enormously increased applicability.

Several emerging issues, such as the use of technology by older adults, the availability of high-capacity Internet access, and support for telemedicine, can be overcome in the near future to increase the benefits of telemedicine.

The question of whether telemedically supervised testing with SARS-CoV-2 Rapid Antigen Tests is non-inferior to the same tests being carried out by trained personnel in test centers is still unanswered.

With this study, the investigators aim to compare and evaluate the reliability and sampling quality of telemedically guided self-performed rapid tests for professional use compared to professional sampling by healthcare personnel.

Our hypothesis is that, applying a strict standard operating procedure (SOP, attached), guided oropharyngeal + nasal (OP+N) self-sampling (GSS) is non-inferior to nasopharyngeal (NP) or OP+N sampling performed by health care professionals (HCP), and that guided OP+N sampling is superior to unsupervised OP+N self-sampling (USS).

PROJECT OBJECTIVES AND DESIGN 2.1 Hypothesis and primary objective

Our hypothesis is that, applying a strict standard operating procedure (SOP, attached), guided oropharyngeal + nasal (OP+N) self-sampling (GSS) is non-inferior to nasopharyngeal (NP) or OP+N sampling performed by health care professionals (HCP), and that guided OP+N sampling is superior to unsupervised OP+N self-sampling (USS).

OP+N GSS is non-inferior to nasopharyngeal (NP) sampling performed by HCP

OP+N GSS is non-inferior to OP+N performed by HCP

OP+N GSS is superior to unsupervised OP+N USS

The investigators are also interested to know if the difference between the sampling techniques is the same depending on the SARS-CoV-2 viral load (low, medium, high).

Another secondary endpoint will be in how many people a correctly executed nasopharyngeal sampling is possible. Due to lack of comfort, deviation of septum, as well as nasal polyps in a small percent of the population, the investigators hypothesize that in a majority of people it is not possible to correctly execute a nasopharyngeal sampling.

2.2 Primary and secondary endpoints

The Ct-value is defined as the number of cycles required for a signal to cross the detection threshold and can be used as a surrogate for sampling quality, as it allows to quantify the amount of material that is being extracted.

Primary endpoints:

Concordance of positive/negative samples in antigen tests with GSS, USS, and HCP-based samples.

Secondary endpoints:

Housekeeping gene Ct comparison based on sampling method between samples based on GSS, USS, or HCP ORF1ab/RdRp-, E-, N-, and S genes Ct value comparison based on sampling method between samples based on GSS, USS, or HCP Qualitative analysis of perceived sampling accuracy established with a short form Detected variant of concern Case report form (CRF) assessing basic demographics and variables of interests as indicated separately in the CRF form Prevalence of variants of concern Immunization status Travel destinations in the passed three months n of people in which a nasopharyngeal sampling is possible correctly (ratio) 2.3 Project design

This is a single-center, randomized, controlled study at a Swiss test station.

2.3.1 Piloting

In order to assess the sampling quality by HCP or telemedically guided self-sampling, Ct values obtained in RT-PCR analysis of a COVID-19 assay, a housekeeping gene can be used for reference.

Hence, for the first part of the study, the investigators will recruit 10 people in which the investigators will perform an OP+N sampling at two-time points, 15 minutes apart, and compare the Ct values of these two values to calculate the standard deviation and see if the produced SD*1.96/√(Sample size) equals the margin of error. Our 95% confidence interval (CI) will be standard deviation (SD)+/- the margin of error.

Alternatively, the investigators will pool confirmed RT-PCRs of two/three swab samples into one and spike them with SARS-CoV-2 standard. Next, the investigators do as many repeats of the same sample on RT-PCR comparing housekeeper and SARS-CoV-2 genes. The advantage here is that the investigators will have controlled starting biological material and the resultant SD / 95% CI will concern only the analytical and laboratory process variability. With the first approach, the investigators will test SD of the swab procurer too, along with the interference coming from the analytical process (lab, instruments, sample storage).

2.3.2. Randomized telemedical and HCP sampling

After giving informed consent by signing the consent form, patients will be randomized to either OP+N GSS - or to OP+N USS.

After performing either procedure, they will continue to be sampled by HCP OP+N and HCP NP.

The investigators will start the assessment with the self-sampling methods in order to reduce bias that could occur if they experience the HCP's sampling.

Written instructions on how to perform a self-test will be provided, representing the instructions that come along with a commercially available rapid test set. An instructional online video tutorial or similar would also account as the latest state of the art.30 However, this has not yet been implemented comprehensively with all available test sets that are currently being distributed across Switzerland.

Furthermore, to avoid bias in the sampling procedure, exclusively one HCP at the testing station will be designated as the study's sampling expert. The HCP will perform the NP and OP+N sampling sequentially in a previously randomized order.

The telemedical guidance will be exclusively done by the same HCP in order to minimize interoperability differences. The standardized telemedical sampling will be conducted at the same test station, in a separate empty room in which a computer will be placed with instructions on how to connect for the telemedical consultation.

During each sampling procedure, the patients will either undergo OP+N GSS or OP+N USS for PCR analysis, as well as for antigenic testing. This means each participant will be sampled a total of six times within 15 minutes from different locations in the upper respiratory tract. Concordance of results between sampling by GSS vs. USS vs. HCPs will be assessed.

As the difference in time between the samplings can influence the Ct value, the sampling process will only be started when the HCP and the telemedical supervisor are ready. The three different samples will be stored in the test station refrigerator between 2°C-8°C before transport.

A grouping of samples will ensure that temperature changes are consistent between samples from the same participant.

PROJECT POPULATION AND STUDY PROCEDURES 3.1 Project population, inclusion and exclusion criteria

All patients, regardless of symptoms, who present themselves at the Test-station SARS-CoV-2 testing will be offered to participate in the study.

Study inclusion criteria; Written informed consent Patients visiting the test-station for a SARS-CoV-2 test Consent to comply with the study protocol Age of 18 or older

List the study exclusion criteria:

Refusal to comply with the study protocol Digital illiteracy (i.e. patients who would never use telemedicine as they do not feel competent enough to use the necessary tools) Not German or English speaking People trained in the use of rapid diagnostic tests (HCP, biologists) will be excluded to reduce bias30

3.2 Recruitment, screening and informed consent procedure All costs for tests performed within the framework of the study will be financed by the study. A payable travel certificate will be issued for unchanged costs. Participation in the study and spending time on it is voluntary, free of charge and at no cost to the study participants. However, each study participant will receive a voucher for free PCR testing at a later date.

Participants will not receive financial compensation for the participation in this study. However, each study participant will receive a voucher for free PCR testing at a later date.

The investigators shall end recruiting either when reaching the necessary sample size or no later than October 30th, 2022.

STATISTICS AND METHODOLOGY 4.1. Statistical analysis plan

4.1.1 Randomization

To ensure allocation concealment, randomization will be performed with a block of 170 in a 1:1 allocation ratio by a web-based independent randomization software (Random Allocation version 1.0). Patients will be randomly assigned to either OP+N GSS or to OP+N USS. Instruction on the assigned procedure will be kept in sealed opaque envelopes labeled with sequential study numbers and opened right before swab-testing.

4.1.2 Sample size

The SD of the mean of Ct values for RT-PCR analysis of multiple samples is not clearly defined in the literature and varies between studies.34,35

If there is truly no difference between the standard and experimental treatment, then 85 patients per group are required to be 90% sure that the lower limit of a one-sided 97.5% confidence interval (or equivalently a 95% two-sided confidence interval) will be above the non-inferiority limit of -3.

We, therefore, estimated a standard error of six that accounts for this variance. In addition, the limit of non-inferiority was set at three according to clinical significance.

Results will be stratified by symptom status, age, and sex.

4.1.3 Hypothesis

Primary outcome

NP HCP vs OP+N HCP H0: μe - μs ≤ -d -> μ(NP HCP ct) - μ(OP+N HCP ct) ≤ -3 H1: μe - μs > -d -> μ(NP HCP ct) - μ(OP+N HCP ct) > -3

OP+N HCP vs OP+N GSS

H0: μe - μs ≤ -d -> μ(OP+N HCP ct) - μ(OP+N GSS ct) ≤ -3 H1: μe - μs > -d -> μ(OP+N HCP ct) - μ(OP+N GSS ct) > -3

OP+N HCP vs OP+N USS

H0: μe - μs ≤ -d -> μ(OP+N HCP ct) - μ(OP+N USS ct) ≤ -3 H1: μe - μs > -d -> μ(OP+N HCP ct) - μ(OP+N USS ct) > -3

Secondary outcome:

We will stratify the primary outcome by viral load (low, medium, high).

4.1.4. Statistical test

A variant of a paired student t test or Wilcoxon test (if non-normal distribution) with exchange of null and alternative (relaxed) hypotheses will be used as a non-inferiority test to assess differences in cycle threshold (Ct, considered as a log2-transformed measure of the amount of viral RNA load) between the NP and OP/N samples (HCP and GSS). Stratification for possible confounders will be done using logistic regression.

In order to show agreement between the approaches and estimate the limits of agreement and those are not too large, different graphical methods, such as Bland Altman diagrams will be used to show agreement between the approaches.

4.2. Handling of missing data Analysis is based on intention-to-treat assumption. Collected data until drop-out will be included for further analysis.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Patients visiting the test-station for a SARS-CoV-2 test
* Consent to comply with the study protocol
* Age of 18 or older

Exclusion Criteria:

* Refusal to comply with the study protocol
* Digital illiteracy (i.e. patients who would never use telemedicine as they do not feel competent enough to use the necessary tools)
* Not German or English speaking
* People trained in the use of rapid diagnostic tests (HCP, biologists) will be excluded to reduce bias

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2022-04-14 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
NP HCP vs OP+N HCP | 5 months
  Concordance of positive/negative samples in antigen tests with nasopharyngeal sampling vs. oropharyngeal + nasal sampling, both performed by health care professionals
OP+N HCP vs OP+N GSS | 5 months
  Concordance of positive/negative samples in antigen tests with oropharyngeal + nasal sampling performed by health care professionals vs. oropharyngeal + nasal sampling telemedically guided self-sampling
OP+N HCP vs OP+N USS | 5 months
  Concordance of positive/negative samples in antigen tests with oropharyngeal + nasal sampling performed by health care professionals vs. unsupervised oropharyngeal + nasal self-sampling (USS)

SECONDARY OUTCOMES:
Housekeeping gene Ct comparison of oropharyngeal + nasal samples between guided self-sampling, unsupervised self-sampling, or sampling performed by health care professionals | 5 months
  Housekeeping gene Ct* comparison of oropharyngeal + nasal samples between guided self-sampling, unsupervised self-sampling, or sampling performed by health care professionals
  *The Ct (cycle threshold) is defined as the number of cycles required for the viral genetic material to be detected above a certain level.
ORF1ab/RdRp-, E-, N-, and S genes Ct value comparison based on sampling method between samples based on GSS, USS, or HCP | 5 months
  ORF1ab/RdRp-, E-, N-, and S genes Ct value comparison based on sampling method between samples based on GSS, USS, or HCP
  Abbreviations:
  ORF1ab/RdRp-, E-, N-, and S genes are different houskeeping genes that serve as a reference level to compare the amount of the viral genetic material The Ct (cycle threshold) is defined as the number of cycles required for the viral genetic material to be detected above a certain level.
  GSS: guided self-sampling USS: unsupervised self-sampling HCP: sampling performed by health care professionals
Qualitative analysis of perceived sampling accuracy | 5 months
  Qualitative analysis of perceived sampling accuracy established with a short form
Detected SARS-CoV-2 variants of concern | 5 months
  The detected SARS-CoV-2 Variants of Interest and Concern (VOC) is recorded. The WHO homepage is consulted for the specification: https://www.who.int/activities/tracking-SARS-CoV-2-variants
CRF assessing basic demographics and variables of interests | 5 months
  Case report form (CRF) assessing basic demographics and variables of interests as indicated separately in the CRF form
Prevalence of variants of concern | 5 months
  Prevalence of each detected variant of concern
Immunization status regarding previous COVID-Vaccinations or previous COVID-19 disease(s) | 5 months
  Type and date of previous previous COVID-vaccinations and COVID-19 diseases basing on positive test results or detected serologic antibodies will be recorded. These facts are requested and verified with the respective patient-specific COVID certificate.
Travel destinations in the passed three months | 5 months
  Travel destinations in the passed three months before the current sampling in the form of countries travelled to and, where appropriate, regions
n of people in which a nasopharyngeal sampling is possible correctly (ratio) | 5 months
  n of people in which a nasopharyngeal sampling is possible correctly (ratio)
  - reason for impossible correct sampling would be anatomical variations of the nose or pathological anatomical conditions

CONTACTS AND LOCATIONS:
Overall Officials: Christian V Eisenring, MD, Principal Investigator — Teststation Praxis Dr. med Bielecki
Locations (1):
- Teststation Praxis Dr. med Bielecki, Olten, Canton of Solothurn, Switzerland

IPD SHARING:
Plan to Share IPD: No
The individual participant data will be entered into REDCap, an online CRF. Access is only possible with a username and password. De-indentified data will be downloaded after study completion and stored for ten years.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-14): https://cdn.clinicaltrials.gov/large-docs/07/NCT05386407/Prot_SAP_000.pdf